CLINICAL TRIAL: NCT04799587
Title: The Use of P6 Acupressure for the Reduction of Intraoperative and Postoperative Nausea and Vomiting in Women Undergoing Cesarean Delivery: a Randomized Trial
Brief Title: Accupressure of P6 to Reduce Nausea During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Feyce M. Peralta, MD, MS, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU#: 00213854
Record Dates: First submitted 2021-02-26; First posted 2021-03-16 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Related; Cesarean Delivery; Nausea; Vomiting
Keywords: Accupressure; Cesarean Delivery; Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: Two group, sham vs actual location of pressure point.
Who Masked: Participant
Masking Description: Participant will not know whether the pressure point is correct or sham location.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P6 Accupressure Group (Active Comparator): The pressure point will be stimulated by the presence of the magnet when positioned properly on the P6 acupressure point. Additional pressure may be applied as desired by the study subject but is not necessary for P6 stimulation.
  Interventions: Other: Magnet at P6
- Sham Pressure Point (Sham Comparator): The sham pressure point (distal to the P6 acupressure point).
  Interventions: Other: Magnet applied to arm not at P6 pressure point.

INTERVENTIONS:
Other: Magnet at P6 — Magnet applied at P6 and attached with adhesive tape. The P6 pressure point is 2 inches proximal to the flexor retinaculum, between the flexor carpi radialis and palmaras longus.
  Arms: P6 Accupressure Group
Other: Magnet applied to arm not at P6 pressure point. — Magnet applied to arm not at P6 pressure point and affixed with adhesive tape.
  Arms: Sham Pressure Point

SUMMARY:
The purpose of this study is to evaluate if the addition of P6 pressure point stimulation as opposed to sham-point stimulation will decrease intraoperative and postoperative nausea and vomiting (IONV and PONV) for patients undergoing non-emergent cesarean delivery. We hypothesize that the addition of stimulation of the P6 pressure point to our institutional current standard of care (phenylephrine infusion, intravenous fluid bolus, and as needed intraoperative ondansetron) will decrease the occurrence of intraoperative emesis.

DETAILED DESCRIPTION:
After obtaining written informed consent from the subject. They were then randomized to either the P6 acupressure or a sham acupressure group. Envelopes containing group assignment information were prepared prior to the start of the study by research personnel not involved in this study. Randomization occurred by selecting a sealed envelope that contained the group assignment, two acupressure 0.09-inch by 0.2-inch diameter devices, and a diagram of where to place the device from a pool of 200 envelopes. The acupressure devices used in this study are also used in clinical practice by Northwestern Medicine Osher Center for Integrative Medicine (Plaster - Accu Band 800 NP Magnets, Japan). Prior to the commencement of the study, the Center for Integrative Medicine acupuncturists educated study personnel on the placement of the devices and the proper patient-initiated stimulation method when the subject began to perceive nausea. Device placement took place in the preoperative room, prior to walking to the operating room for the surgical procedure, by research personnel not involved in the clinical care of study subjects. In the P6 acupressure group, the devices were placed two inches proximal to the flexor retinaculum, between the flexor carpi radialis and palmaras longus bilaterally. The small protrusion on the device was placed on the skin and held in place using an adhesive sticker at the stimulation point. In the sham acupressure group, the devices were placed distal and lateral to the P6 acupoint site, like in prior studies comparing the effectiveness of P6 acupressure to sham. This method of sham acupoint placement when compared to P6 acupoint placement has shown superiority of the P6 acupoint placement in 70% of studies that have used this point for sham.15 The devices are designed to maintain pressure at the point of placement without additional force applied. Research personnel also instructed subjects to apply additional pressure at the acupressure site for a period of 30 s-2 min if they perceived nausea. Subjects were then taken to the operating room where they received neuraxial anesthesia consisting of either a spinal anesthetic dosed with hyperbaric bupivacaine 12 mg plus fentanyl 15 mcg and morphine 150 mcg, or a combined spinal epidural with the same intrathecal dosing per institutional standard practice. Co-loading with a crystalloid solution occurred upon the start of the neuraxial procedure, and a phenylephrine infusion was started immediately after the cerebrospinal fluid was obtained. Maternal hypotension was defined as a systolic blood pressure less than 100 mmHg, mean arterial pressure less than 65 mmHg, or mean arterial pressure less than 20% of the baseline mean arterial pressure. The baseline blood pressure was considered the average value of three blood pressure readings obtained by the nursing staff in the preoperative area. Subjects were asked to report any nausea, retching, or vomiting to the anesthesia care team. In addition, the anesthesia provider asked the study subject about nausea or vomiting at intervals corresponding to events that are associated with a greater prevalence of nausea and vomiting (e.g. neuraxial dose administration, uterine exteriorization, and following uterotonic administration) as well as when the anesthesia provider observed the subject massaging the acupressure point. After the first complaint of nausea, subjects were encouraged to apply additional pressure to the devices, an intravenous (IV) fluid bolus was administered, and phenylephrine or ephedrine was administered by IV bolus and/or by increasing the infusion rate of phenylephrine if hypotension was present. At the second complaint of nausea or emesis, study subjects were again encouraged to apply additional pressure on the devices. Following delivery of the fetus, ondansetron 8 mg IV and dexamethasone 8 mg IV were administered. If intraoperative nausea and/or vomiting continued, study subjects were again encouraged to apply additional acupressure. If this was ineffective, prochlorperazine, promethazine, metoclopramide, fentanyl, or propofol were administered at the anesthesiologist's discretion. If these antiemetic agents were ineffective, the anesthesiologist could provide additional medications.

Routine postoperative orders, including antiemetic medications as needed, were placed by the anesthesiology team for postpartum use per our institution's current standard of care. Postoperative medications were administered and documented by the nursing staff. Study subjects were also encouraged to use additional acupressure as needed throughout their postoperative course, for up to 48 h or until discharge, whichever came first. A study team member replaced devices that were lost or removed the device if the study subject requested it. Prior to discharge, subjects were visited by study personnel and asked to complete a survey asking them to describe the incidence, duration, and severity of nausea and vomiting, interference of nausea/vomiting with the ability to care for themselves, and their rating and satisfaction of the acupressure therapy.

Baseline data collected were age, weight, height, body mass index, American Society of Anesthesiologists physical status classification, race, ethnicity, history of nausea and vomiting, parity, and the number of prior cesarean delivery. Intraoperative data included the type of neuraxial anesthesia, initial blood pressure in the operating room, the lowest recorded blood pressure intraoperatively, total vasopressor use (expressed as phenylephrine equivalents),18 the number of hypotensive episodes, crystalloid administered, and duration of anesthesia. Intraoperative nausea and vomiting outcomes included the number of subjects with nausea and/or vomiting, the number of emesis episodes, and the need for rescue antiemetic administration in the operating room. Post delivery emesis and antiemetic treatments were recorded in the post anesthesia care unit (PACU) in 0-24 h and 24-48 h periods. Study subject questionnaires were collected at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* English-speaking
* Pregnant patients presenting for scheduled cesarean delivery of a full-term fetus (>37 weeks' gestation)
* Patients scheduled as ERAC
* Parturients undergoing spinal anesthesia

Exclusion Criteria:

* Patients requiring emergent delivery,
* Fetal demise
* Patients with adhesive allergy/sensitivity
* Patients with allergy/sensitivity to nickel,
* Patients with inability to consent,
* Patients with known abnormal placentation
* Patients with pacemakers/defibrillators
* Patients with positive COVID-19 tests

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy
Enrollment: 200 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feyce Peralta, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balki M, Carvalho JC. Intraoperative nausea and vomiting during cesarean section under regional anesthesia. Int J Obstet Anesth. 2005 Jul;14(3):230-41. doi: 10.1016/j.ijoa.2004.12.004. PMID 15935649
- [Background] Chooi C, Cox JJ, Lumb RS, Middleton P, Chemali M, Emmett RS, Simmons SW, Cyna AM. Techniques for preventing hypotension during spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2017 Aug 4;8(8):CD002251. doi: 10.1002/14651858.CD002251.pub3. PMID 28976555
- [Background] Ho CM, Tsai HJ, Chan KH, Tsai SK. P6 acupressure does not prevent emesis during spinal anesthesia for cesarean delivery. Anesth Analg. 2006 Mar;102(3):900-3. doi: 10.1213/01.ane.0000195553.82409.00. PMID 16492848
- [Background] Albooghobeish M, Mohtadi A, Saidkhani V, Fallah H, Behaein K, Nesionpour S, Nikbakht R. Comparison Between Effects of Acupuncture and Metoclopramide on Postoperative Nausea and Vomiting after Gynaecological Laparoscopy: A Randomized Controlled Trial. Anesth Pain Med. 2017 Aug 22;7(5):e12876. doi: 10.5812/aapm.12876. eCollection 2017 Oct. PMID 29696109
- [Background] Lee A, Fan LT. Stimulation of the wrist acupuncture point P6 for preventing postoperative nausea and vomiting. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD003281. doi: 10.1002/14651858.CD003281.pub3. PMID 19370583
- [Background] Matthews A, Haas DM, O'Mathuna DP, Dowswell T. Interventions for nausea and vomiting in early pregnancy. Cochrane Database Syst Rev. 2015 Sep 8;2015(9):CD007575. doi: 10.1002/14651858.CD007575.pub4. PMID 26348534
- [Background] Allen TK, Habib AS. P6 stimulation for the prevention of nausea and vomiting associated with cesarean delivery under neuraxial anesthesia: a systematic review of randomized controlled trials. Anesth Analg. 2008 Oct;107(4):1308-12. doi: 10.1213/ane.0b013e31816d1864. PMID 18806045
- [Background] Habib AS, Itchon-Ramos N, Phillips-Bute BG, Gan TJ; Duke Women's Anesthesia (DWA) Research Group. Transcutaneous acupoint electrical stimulation with the ReliefBand for the prevention of nausea and vomiting during and after cesarean delivery under spinal anesthesia. Anesth Analg. 2006 Feb;102(2):581-4. doi: 10.1213/01.ane.0000189217.19600.5c. PMID 16428565
- [Background] El-Deeb AM, Ahmady MS. Effect of acupuncture on nausea and/or vomiting during and after cesarean section in comparison with ondansetron. J Anesth. 2011 Oct;25(5):698-703. doi: 10.1007/s00540-011-1198-0. Epub 2011 Jul 15. PMID 21761206
- [Background] Tan JY, Suen LK, Wang T, Molassiotis A. Sham Acupressure Controls Used in Randomized Controlled Trials: A Systematic Review and Critique. PLoS One. 2015 Jul 15;10(7):e0132989. doi: 10.1371/journal.pone.0132989. eCollection 2015. PMID 26177378
- [Background] Wengritzky R, Mettho T, Myles PS, Burke J, Kakos A. Development and validation of a postoperative nausea and vomiting intensity scale. Br J Anaesth. 2010 Feb;104(2):158-66. doi: 10.1093/bja/aep370. Epub 2009 Dec 26. PMID 20037151
- [Background] Boogaerts JG, Vanacker E, Seidel L, Albert A, Bardiau FM. Assessment of postoperative nausea using a visual analogue scale. Acta Anaesthesiol Scand. 2000 Apr;44(4):470-4. doi: 10.1034/j.1399-6576.2000.440420.x. PMID 10757584
- [Background] Sheldon RR, Loughren MJ, Marenco CW, Winters JR, Bingham JR, Martin MJ, Eckert MJ, Burney RO. Microdermal Implants Show No Effect on Surrounding Tissue During Surgery With Electrocautery. J Surg Res. 2019 Sep;241:72-77. doi: 10.1016/j.jss.2019.03.039. Epub 2019 Apr 19. PMID 31009888
- [Background] A DM, A K. Effect of acupressure on post-operative nausea and vomiting in cesarean section: a randomised controlled trial. J Clin Diagn Res. 2013 Oct;7(10):2247-9. doi: 10.7860/JCDR/2013/5702.3485. Epub 2013 Oct 5. PMID 24298488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 200 consented 1 dropped out in the P6 treatment group.
Period: Overall Study
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Started | 100 | 100
Completed (P6 group 1 subject withdrew consent to participate.) | 100 | 99
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Pressure Point | P6 Accupressure Group | Total
Number analyzed (Participants) | 100 | 99 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 99 | 199
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.6 (4.5) | 35.3 (4.8) | 35 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 99 | 199
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 20 | 46
  Not Hispanic or Latino | 74 | 79 | 153
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 16 | 26
  White | 79 | 76 | 155
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 100 | 99 | 199
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 163 (7.5) | 164 (7.5) | 163 (7.5)
Weight (kg) [Mean (Standard Deviation); unit: Kilograms] | 86 (19) | 89 (18) | 87 (18)
Body Mass Index (kg/m^2) [Median (Inter-Quartile Range); unit: kg/m^2] | 31.6 [28.1 to 37.3] | 31.4 [27.9 to 37.3] | 31.5 [27.9 to 37.3]
American Society of Anesthesiology (ASA) physical status n [Count of Participants; unit: Participants] — ASA (American Society of Anesthesiologists) physical status classification system is a tool used to assess a patient's overall health and risk of complications during surgery. It grades patients from ASA 1 (healthy) to ASA 5 (moribund).
  Participants
    ASA 2 | 74 | 81 | 155
    ASA 3 | 26 | 18 | 44
Parity [Count of Participants; unit: Participants]
  0 | 15 | 27 | 42
  1 | 55 | 46 | 101
  2 | 23 | 18 | 41
  3 | 7 | 8 | 15
Prior cesarean delivery (n) [Count of Participants; unit: Participants]
  No prior cesarean delivery | 25 | 31 | 56
  Yes, previous cesarean delivery | 75 | 68 | 143
Type of neuraxial anesthesia [Count of Participants; unit: Participants]
  Spinal | 93 | 86 | 179
  Combined spinal epidural | 7 | 13 | 20
Initial BP in operating room (mmHg) [Median (Inter-Quartile Range); unit: mmHg]
  Systolic | 136 [124 to 150] | 134 [121 to 151] | 135 [121 to 151]
  Diastolic | 82 [74 to 88] | 79 [72 to 90] | 80 [72 to 90]
History of nausea/vomiting [Count of Participants; unit: Participants]
  No | 55 | 50 | 105
  Yes | 45 | 49 | 94

OUTCOME MEASURES:

1. Primary Outcome: Presence of Intraoperative Vomiting
Description: Presence of intraoperative vomiting during scheduled cesarean delivery (intraoperative period).
Time Frame: Intraoperative Period
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 100 | 99
Participants | 17 | 17
Statistical Analysis 1: Comparison: Sham Pressure Point vs P6 Accupressure Group; The incidence of nausea and vomiting and the number of episodes between the P6 acupressure and sham acupressure groups were compared using a chi-square statistic (nominal data) or the Wilcoxon test (continuous data); Test type: Superiority — Sample size for the study was determined by assuming a baseline rate of 33% of IONV and that there will be a relative decrease of 50% in the group that receives P6 acupressure during CD. A two-sided Fisher's Exact Test, with a significance level of 0.05, group sizes of 98 are needed to achieve 80% power to detect a difference between the group proportions of 0.18. Group sizes were rounded up to 100. Statistical analyses were two-sided, and a P<0.05 was required to reject the null hypothesis; p = .94, Chi-squared

2. Primary Outcome: Presence of Intraoperative Nausea
Description: Presence of intraoperative nausea during scheduled cesarean delivery (intraoperative period).
Time Frame: Intraoperative period
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 100 | 99
Participants | 57 | 56
Statistical Analysis 1: Comparison: Sham Pressure Point vs P6 Accupressure Group; The sample size for the study was determined by assuming a baseline rate of 33% of intraoperative nausea and vomiting and that there will be a relative decrease of 50% in the group that receives P6 acupressure during CD.20 Using a two-sided Fisher's Exact Test, with a significance level of 0.05, group sizes of 98 are needed to achieve 80% power to detect a difference between the group proportions of 0.18. Group sizes were rounded up to 100; Test type: Superiority; p = .95, Chi-squared

3. Secondary Outcome: Number of Emesis Episodes in the Intraoperative Period Period
Description: The number of emesis episodes during the cesarean section intraoperative period.
Time Frame: Intraoperative period
Population: Reported number of emesis episodes based on number of subjects who experienced emesis .
  17 in sham group and 17 in the P6 acupressure group.
Measure: Median (Inter-Quartile Range); unit: Emesis episodes
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 17 | 17
Emesis episodes | 2 [1 to 4] | 2 [1 to 4]

4. Secondary Outcome: Number of Rescue Antiemetic Doses Administered for the Treatment of Intraoperative Nausea and Vomiting
Description: Reported total number (count) of rescue antiemetics administered per group during the intraoperative period. Rescue antiemetics are defined as the use of intravenous administered prochlorperazine, promethazine, or metoclopramide.
Time Frame: Intraoperative period
Population: Number of antiemetic and/or anti-nausea medications administered in the intraoperative period.
Measure: Number; unit: Number of antiemetics per group
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 100 | 99
Number of antiemetics per group | 10 | 10

5. Other Pre Specified Outcome: The Number of Emesis From Post Anesthesia Care Unit to Discharge.
Description: Reported total number (count) of emesis episodes per group from admission to the post anesthesia care unit after the operative procedure to discharge from the hospital.
Time Frame: 96 hours
Measure: Number; unit: Emesis episodes
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 100 | 99
Emesis episodes | 17 | 13

6. Other Pre Specified Outcome: Antiemetic Medication Administered From the PACU Through Discharge
Description: The number(count) of antiemetic medication administered per group in the post anesthesia care unit through discharge from the hospital
Time Frame: 96 hours
Measure: Number; unit: Doses administered
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 100 | 99
Doses administered | 27 | 30

7. Other Pre Specified Outcome: Patient Questionnaire: Have You Experienced Dry Retching or Vomiting
Description: Patient recovery questionnaire administered prior to discharge from the hospital. Have you experienced dry retching or vomiting?
Time Frame: 96 Hours
Population: 73 in the sham group and 74 in the P6 group completed the survey question
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 73 | 74
Participants
  Has experienced dry retching | 3 | 10
  Has experienced vomiting | 20 | 20

8. Other Pre Specified Outcome: Patient Questionnaire: Number of Times Vomited
Description: Patient recovery questionnaire administered prior to discharge from the hospital. (of those who indicated vomiting) How many times did you vomit.
Time Frame: 96 Hours
Population: 73 in the sham group and 74 in the P6 group completed the survey question
Measure: Median (Inter-Quartile Range); unit: Vomit episodes
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 73 | 74
Vomit episodes | 2 [1 to 4] | 2 [1 to 4]

9. Other Pre Specified Outcome: Number of Participants With Nausea
Description: Patient recovery questionnaire administered prior to discharge from the hospital. Have you experienced nausea?
Time Frame: 96 Hours
Population: 73 in the sham group and 74 in the P6 group completed the survey question
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 73 | 74
Participants | 51 | 53

10. Other Pre Specified Outcome: Patient Questionnaire: Describe the Pattern of Your Nausea?
Description: Patient recovery questionnaire administered prior to discharge from the hospital. (of those who had nausea)Describe the pattern of your nausea (2 choices).
Time Frame: 96 Hours
Population: 73 in the sham group and 74 in the P6 group completed the survey question. 51 in the sham group and 53 in the P6 group reported nausea.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 51 | 53
Participants
  Nausea comes and goes | 40 | 44
  Nausea is constant | 5 | 2
  No response | 6 | 7

11. Other Pre Specified Outcome: Patient Questionnaire: Did the Nausea Interfere With You Ability to Care for Yourself?
Description: Patient recovery questionnaire administered prior to discharge from the hospital. (of those who had nausea) How did the nausea interfere with your ability to care for yourself.
Time Frame: 96 Hours
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 51 | 53
Participants
  No interference | 36 | 34
  A little interference | 11 | 11
  Some of the time | 1 | 2
  Most of the time | 3 | 4
  No response | 0 | 2

12. Other Pre Specified Outcome: Patient Questionnaire: Duration of Nausea.
Description: Patient recovery questionnaire administered prior to discharge from the hospital. (of those who had nausea) How many hours did the nausea last.
Time Frame: 96 Hours
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 51 | 53
Hours | 2 [.5 to 14] | 4 [2 to 8]

13. Other Pre Specified Outcome: Patient Questionnaire: Severity of Nausea.
Description: Patient recovery questionnaire administered prior to discharge from the hospital. (of those who had nausea).Severity of nausea based on a 0 (none) -100 (very severe).
Time Frame: 96 Hours
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: score on a scale (0 good-100 severe)
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 51 | 53
score on a scale (0 good-100 severe)
  Highest level of nausea | 50 [18 to 70] | 63 [29 to 78]
  Lowest level of nausea | 4 [0 to 17] | 4 [0 to 23]

14. Other Pre Specified Outcome: Patient Questionnaire: Do You Think the Magnet Improves Nausea?
Description: Patient recovery questionnaire administered prior to discharge from the hospital. Does the magnet improve nausea response yes or no.
Time Frame: 96 Hours
Population: Please note 62 in the sham group and 64 in the P6 group completed this survey question.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 62 | 64
Participants
  Improves nausea (yes) | 23 | 25
  Does not improve nausea (no) | 39 | 39

15. Other Pre Specified Outcome: Patient Questionnaire: Do You Think the Magnet Improves Vomiting?
Description: Patient recovery questionnaire administered prior to discharge from the hospital. Does the magnet improve vomiting response yes or no.
Time Frame: 96 Hours
Population: Please not that 60 in the sham group and 62 in the P6 group completed the survey question.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 60 | 62
Participants
  Improves vomiting (yes) | 15 | 19
  Does not improve vomiting (no) | 45 | 43

16. Other Pre Specified Outcome: Patient Questionnaire: Are You Satisfied With Acupressure?
Description: Patient recovery questionnaire administered prior to discharge from the hospital. Are you satisfied with acupressure response yes or no.
Time Frame: 96 Hours
Population: 61 in the sham group and 65 in the P6 group completed the survey question.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 61 | 65
Participants
  Satisfied with acupressure (yes) | 29 | 33
  Not satisfied with acupressure (no) | 32 | 32

17. Other Pre Specified Outcome: Intraoperative Lowest BP (mmHg)
Description: Lowest systolic and diastolic blood pressure during the intraoperative period.
Time Frame: Intraoperative period
Measure: Mean (Inter-Quartile Range); unit: mm/Hg
Arm/Group | P6 Accupressure Group | Sham Pressure Point
Number analyzed (Participants) | 100 | 99
mm/Hg
  Systolic Blood Pressure | 116 [106 to 124] | 111 [105 to 121]
  Diastolic Blood Pressure | 61 [56 to 69] | 60 [56 to 69]

18. Other Pre Specified Outcome: Intraoperative Total Vasopressor (VPE) [1]
Description: Measure Description: Total vasopressor units expressed as phenylephrine units using an 80:1 ratio for ephedrine in micrograms.
Time Frame: Intraoperative period
Measure: Median (Inter-Quartile Range); unit: micrograms
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 100 | 99
micrograms | 2052 [1288 to 2918] | 2190 [1550 to 2950]

19. Other Pre Specified Outcome: Intraoperative Hypotension Episodes (n)
Description: Number of hypotension episodes experienced during the intraoperative period.
Time Frame: Intraoperative
Measure: Median (Inter-Quartile Range); unit: Hypotension episodes
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 100 | 99
Hypotension episodes | 1 [0 to 2] | 1 [0 to 2]

20. Other Pre Specified Outcome: Intraoperative Crystalloid Co-load (mL)
Description: Amount of crystalloid fluids given as a co-load in milliliters during the intraoperative period.
Time Frame: Intraoperative period
Measure: Median (Inter-Quartile Range); unit: Milliliters
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 100 | 99
Milliliters | 500 [300 to 600] | 500 [300 to 600]

21. Other Pre Specified Outcome: Intraoperative Fluids Administered (mL)
Description: Total number of milliliters of fluids administered during the intraoperative period.
Time Frame: Intraoperative
Measure: Median (Inter-Quartile Range); unit: Milliliters
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 100 | 99
Milliliters | 2000 [1600 to 2175] | 1800 [1500 to 2100]

22. Other Pre Specified Outcome: Duration of Intraoperative Anesthesia (Min)
Description: Duration of administration of intraoperative anesthesia in minutes.
Time Frame: Intraoperative period
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Sham Pressure Point | P6 Accupressure Group
Number analyzed (Participants) | 100 | 99
Minutes | 81 [70 to 98] | 81 [73 to 103]

ADVERSE EVENTS:
Time Frame: 72 Hours
Description: Adverse events were collected on a survey provided to the participant up to 72 hours after delivery.
Arm/Group | Sham Pressure Point | P6 Accupressure Group
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/99
Other Adverse Events (participants affected / at risk) | 57/100 | 56/99
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Pressure Point (N=100) | P6 Accupressure Group (N=99)
Nausea (Gastrointestinal disorders) | 57 (57) | 56 (56) — Experienced nausea during the cesarean section operative period
Emesis during operative period (Gastrointestinal disorders) | 17 (43) | 17 (33) — Emesis during the cesarean section procedure.
Emesis in post anesthesia care unit (Gastrointestinal disorders) | 4 (4) | 9 (9) — Emesis post operative in the post anesthesia care unit
Emesis (floor) (Gastrointestinal disorders) | 17 (17) | 13 (13) — Emesis admission to hospital room after operative procedure to 24 hours post operative

LIMITATIONS AND CAVEATS:
* Our study was underpowered to observe a difference between the groups at the rates of IONV observed.
* Could be an element of patient bias and skepticism among Western women as to the effectiveness of non-pharmacologic therapy for the treatment of nausea and vomiting.
* The chosen dose of intrathecal dose of morphine 150 mcg used in this study is higher than that recommended in the PROSPECT guidelines.
* Uterine exteriorization is routinely performed in our practice, could increase IONV.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT04799587/Prot_SAP_000.pdf